CLINICAL TRIAL: NCT00423228
Title: A Randomised, Double-blind, Double-dummy, Oral Donepezil Controlled Study on the Safety and Efficacy of Repeated Monthly Subcutaneous Injections of a Sustained-release Implant of ZT 1 in Patients With Moderate Alzheimer's Disease
Brief Title: Efficacy Study of a ZT-1 Implant in Patients Suffering From Alzheimer's Disease
Acronym: BRAINz
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DEB-ZTSR-201; EUDRACT no. 2006-005161-18
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Moderate Alzheimer's Disease
Keywords: Alzheimer's disease; cognitive impairment; cholinesterase inhibitors; sustained-release implants; long acting treatment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ZT-1 (Experimental): ZT-1 (investigational product)
  Interventions: Drug: ZT-1
- Donepezil (Active Comparator): Donepezil
  Interventions: Drug: Donepezil

INTERVENTIONS:
Drug: ZT-1 — Patients in the ZT-1 treatment group will receive ZT 1-1 mg capsules administered p.o. daily during the first month of treatment, followed by ZT-1 implants (9 mg) administered s.c. during the second month of treatment, followed by ZT-1 implants (12 mg) administered s.c. every 4 weeks during months 3 to 6 of treatment. Patients in the ZT-1 treatment group will receive dummy donepezil capsules during months 2 to 6 of the treatment period.
  Arms: ZT-1
Drug: Donepezil — Patients in the donepezil treatment group will receive donepezil 5 mg capsules administered p.o. during the first month of treatment, followed by donepezil 10 mg/day during months 2 to 6 of the treatment period. Patients in the donepezil treatment group will also receive s.c. injections of dummy ZT 1 implants every 4 weeks during months 2 to 6 of the treatment period.
  Other Names: Aricept
  Arms: Donepezil

SUMMARY:
Alzheimer's disease is characterised by memory loss and difficulties with thinking. These problems may be due to a deficiency in a brain chemical called acetylcholine. Acetylcholine helps transmit messages between nerve cells. Acetylcholine is degraded by an enzyme called "acetylcholinesterase". ZT-1 is a new drug derived from a plant extract already used in China for memory disorders, which blocks the action of the enzyme and restores adequate levels of acetylcholine.

This study will test the safety and efficacy of ZT-1 in the treatment of patients with Alzheimer's disease.

BRAINz stands for Better Recollection for Alzheimer's patients with the Implant of ZT-1.

DETAILED DESCRIPTION:
This is a multicenter, randomised, double-blind, double-dummy, oral donepezil controlled study on the safety and efficacy of repeated monthly s.c. injections of a sustained-release implant of ZT 1 in patients with moderate Alzheimer's Disease.

The study enrolls patients aged >50 years, with moderate AD with a MMSE score at study screening ≥14 and ≤22. The study aims to recruit 128 patients.

The study is divided into 3 periods:

1. A screening period
2. A 6-month treatment period, consisting of one month of titration with an oral medication and 5 months of treatment with an implant administered under the skin every 4 weeks. Oral treatment will be maintained throughout the treatment phase
3. A 2 week follow-up period.

Patients will be randomized in a 1:1 ratio to one of 2 groups: the ZT-1 (investigational product) treatment group or the donepezil (active comparator) treatment group.

The study comprises a total of 11 visits including screening and follow-up. An additional visit for PK/PD assessment is scheduled in about 10% of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of moderately severe probable AD, diagnosed according to the DSM-IV and the NINCDS-ADRDA criteria;
2. MMSE score ≥ 14 and ≤ 22;
3. Male/female patient aged > 50 years; female patients should be of no child-bearing potential or postmenopausal (at least one year after last menses);
4. Body mass index (BMI) between 18 and 29 kg/m2 inclusive;
5. Has a caregiver, is living at home or in an assisted living facility, is able to attend ambulatory study visits;
6. Naïve to donepezil;
7. Has discontinued another AChEI and/or memantine at least 3 months prior to study visit 2 (Day 1);
8. Has a CT or MRI scan excluding another structural brain disease and supporting diagnosis of AD; CT or MRI scan must have been performed within 6 months prior to study visit 2 (Day 1, baseline);
9. Fluent in English (mother tongue or working language);
10. Able to communicate well with the Investigator;
11. Physically able to carry out functional tasks;
12. Has given written informed consent together with the caregiver.

Exclusion Criteria:

1. Presence of any disabling, severe or life-threatening disease (cardiac, respiratory, gastro-intestinal, neurological, epileptic, psychiatric, infectious, bone, endocrinologic);
2. Inability to discontinue at least 2 weeks prior to visit 2 (Day 1) (or within 5 drug half-lives, whichever is longer) any medication listed as prohibited;
3. Proven or clinically suspected other type of dementia such as vascular dementia, post-traumatic dementia, fronto-temporal dementia, dementia associated with Parkinson's Disease, infectious disease HIV, syphilis), folate or vitamin B12 deficiency, hypothyroidism etc.;
4. Significant liver impairment with ASAT, ALAT >=3x the upper normal limit at screening;
5. Significant kidney impairment with serum creatinine >=2x the upper normal limit at screening;
6. Presence of cardiac rhythm disorder, in particular bradycardia (< 60 bpm), conduction abnormalities such as AV block; presence of active ischaemia (such as unstable angina pectoris) or recent myocardial infarction, QT interval ≥ 450 msec at screening, QRS complex ≥ 110 msec at screening (ECG must be within normal limits at screening);
7. Uncontrolled arterial hypertension i.e. patients with systolic blood pressure (BP) >=160 mmHg and/or diastolic >=100 mmHg, at screening despite regular medication;
8. Uncontrolled arterial hypotension, i.e. patients with systolic BP ≤ 100 mmHg and/or presenting a fall of systolic BP ≥ 20 mmHg or a fall of diastolic BP >=10 mmHg after the 2 min Schellong test at screening;
9. Any concomitant disorder or resultant therapy that is likely to interfere with patient compliance or his/her participation to the study;
10. Participation in another study with an experimental drug within 3 months before study visit 2 (Day 1, baseline) or within 5 drug half-lives of the investigational drug (whichever is the longer);
11. Known peripheral cholinergic intolerance, i.e. with previously prescribed AChEI(s);
12. Known hypersensitivity to any of the test materials or related compounds, including lactose, present in the donepezil and placebo capsules;
13. Known active use of recreational drug or alcohol dependence, current alcohol abuse;
14. Inability to comply fully with the protocol;
15. Patients who, in the opinion of the Investigator, are considered unsuitable for any other reason.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2007-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Change in the MMSE score from baseline to week 25 | baseline to week 25

SECONDARY OUTCOMES:
Responder rate as defined by at least 2 points improvement in the MMSE score; | baseline to week 25
Change on the ADAS-Cog 11 items subscale; | baseline to week 25
Change in the NPI-Q; | baseline to week 25
Change on the IADL scale; | baseline to week 25
Patient's convenience questionnaire. | baseline to week 25

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Tamches, MD, Study Director — Debiopharm SA
Locations (28):
- Australia (9):
  - Central Coast Neuroscience Research, East Gosford, New South Wales
  - Hornsby-Kuring-gai Health Service, Hornsby, New South Wales
  - Southern Neurology, Kogarah, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Queen Elizabeth Hospital, Woodville, South Australia
  - St George's Hospital, Kew, Victoria
  - Austin Health Repatriation Hospital, West Heidelberg, Victoria
  - Hollywood Specialist Centre, Nedlands (Perth), Western Australia
- Canada (11):
  - Calgary West Medical Centre, Calgary, Alberta
  - Castledowns Medicentre, Edmonton, Alberta
  - Saibal Nandy Professional Corporation, Medicine Hat, Alberta
  - Parkwood Hospital, London, Ontario
  - Toronto Memory Program, Toronto, Ontario
  - Gerontion Research Inc., Toronto, Ontario
  - Neuro Rive-Sud, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - The Medical Arts Health Research Group, Kelowna
  - Douglas Hospital Research Center, Montreal
  - The Medical Arts Health Research Group, Penticton
- United Kingdom (8):
  - OPMHS, Crowborough, East Sussex
  - Camden and Islington Mental Health Trust, London, London
  - Glasgow Memory Clinic, Glasgow, Scotland
  - Llandough Hospital, Penarth, Wales
  - Royal Blackburn Hospital, Blackburn
  - North Manchester General Hospital, Manchester
  - New Castle General Hospital, Newcastle upon Tyne
  - MARC - Moorgreen Hospital, Southampton

REFERENCES:
- [Background] Wilkinson D, Roughan L. The BRAINz trial: a novel approach to acetylcholinesterase-inhibitor treatment for Alzheimer's disease. Future Neurol 2(4):379-382,2007.
- See also: Sponsor of the Study — http://www.debiopharm.com
- See also: Alzheimer's Disease Education and Referral (ADEAR) Center — http://www.alzheimers.org